CLINICAL TRIAL: NCT03113994
Title: The Efficacy and Safety of Rosuvastatin for Modifying Bone Mass and Cardiometabolic Disease Outcomes
Brief Title: Statin Monotherapy for Treatment of Endocrine Metabolic Disease Risk
Acronym: RoBaCO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. B. Catharine. Craven (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Toronto Rehabilitation Institute (Other); University Health Network, Toronto (Other); University of Miami (Other); Rick Hansen Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. B. Catharine. Craven, Clinician Scientist/Principal Investigator, Toronto Rehabilitation Institute
Organization: Toronto Rehabilitation Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-350642
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries; Osteoporosis; Metabolic Syndrome
Keywords: Spinal Cord Injury; Osteoporosis; Cardiometabolic Syndrome
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis; Metabolic Syndrome | interventions — Rosuvastatin Calcium; coenzyme Q10; Calcium Carbonate; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin Calcium; Dietary Supplement: Coenzyme Q10; Dietary Supplement: Calcium Carbonate; Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet; Dietary Supplement: Coenzyme Q10; Dietary Supplement: Calcium Carbonate; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Rosuvastatin Calcium — 10mg Rosuvastatin, daily for 12 months
  Arms: Rosuvastatin
Drug: Placebo Oral Tablet — Placebo, daily for 12 months
  Arms: Placebo
Dietary Supplement: Coenzyme Q10 — 100mg CoQ10, daily for 12 months
Dietary Supplement: Calcium Carbonate — 1250mg Calcium Carbonate, daily for 12 months
Dietary Supplement: Vitamin D — 2000IU Vitamin D, daily for 12 months

SUMMARY:
Rationale: After having a spinal cord injury (SCI), people develop changes in their body composition that influences their long-term health. Individuals with paralysis after SCI will have large declines in their bone density ant increases in fat mass which increases their risk of fracture and heart disease. Therapies to prevent SCI-related changes in body composition and their health effects are needed. Drugs known as "statins" used often to reduce high cholesterol, may help to reduce bone loss and inflammation.

Hypothesis: Among adults with SCI for a long time, treatment with a drug named Rosuvastatin or a sugar pill, with supplements (coenzyme Q10, calcium and vitamin D), for twelve months can decrease their endocrine metabolic disease risk by increasing bone density and reducing inflammation.

Study Design: A clinical trial will be conducted in Toronto, Ontario and Miami, Florida. Subjects will get statin therapy or placebo (sugar pill) by chance. Study subjects and research staff will not know whether they are taking the study drug or a sugar pill until after the study

Subjects: Fifty-four adults (age 18-60 years) with a long-term SCI and no movement below their level of injury.

Treatment: Subjects will be prescribed Rosuvastatin 10 mg daily or a sugar pill. In addition, all subjects will receive 100 mg of Co-Q10 daily, calcium carbonate 1250 mg and, vitamin D 2,000 IU once a day.

Data Collected: Subjects' bone density will be collected at the start and end of the study. Change in bone density between the two groups will be compared to see if one is better. Blood samples will be collected quarterly to make sure subjects are safe and do not develop problems with their liver or muscles and to measure the effects of the study drugs on inflammation throughout the body.

Clinical Implications: Statins may be safe and effective therapy for adults living with SCI who are at increased risk of endocrine metabolic disease as they age.

DETAILED DESCRIPTION:
Rationale: Individuals with motor-complete spinal cord injury (SCI) undergo dramatic changes in body composition in the first 18 months post-injury, including declines in bone mineral density (BMD) that increase lower-extremity fragility fracture risk, and increases in fat mass that increase cardio-metabolic disease (CMD) risk. While statins are an effective treatment for dyslipidemia, research evidence suggests additional pleiotropic effects on bone through promotion of osteogenesis, suppression of osteoblast apoptosis, and inhibition of osteoclastogenesis. There are currently no effective therapies to treat sublesional osteoporosis (SLOP) and reduce the risk of fragility fractures in individuals with SCI.

Hypothesis: Twelve months of statin therapy with concurrent coenzyme Q10 (CoQ10), to reduce risk of statin neuromyotoxicity, and standard care (calcium 1250mg OD and vitamin D3 2000IU OD) will be superior to placebo with CoQ10 and standard care, for augmenting knee region BMD and reducing inflammatory stress (hs-CRP), thereby reducing endocrine metabolic disease risk.

Objective: To determine the safety and efficacy of statin therapy for augmenting distal femoral BMD among adults with chronic motor-complete SCI in Toronto, Ontario and Miami, Florida.

Study Design: Multi-centre, double-blind, randomized controlled Phase II safety and efficacy trial.

Subjects: Consenting men and premenopausal women (N=54, age 18-60 yrs) with chronic (≥2 years) spinal cord injury with a neurological level between C1-T10 and an AIS category of A/B.

Intervention: Rosuvastatin 10 mg po daily at night versus placebo for 12 months. All subjects will receive osteoporosis standard care (calcium carbonate 1250mg po daily and vitamin D3 2000 IU po daily) to maintain bone mass and CoQ10 100mg po daily to prevent statin-induced myopathy.

Outcomes: Primary safety outcomes: i) establish the safety of rosuvastatin in chronic SCI by reporting the frequency of myotoxicity and type II diabetes onset; ii) frequency and mean duration of liver transaminase elevations in the rosuvastatin and placebo groups. Primary efficacy outcome: measure the mean between group absolute changes in distal femur areal BMD (aBMD, g/cm2) from baseline to one year. Secondary efficacy outcomes: will examine the mean absolute changes from baseline in: i) volumetric BMD (vBMD, g/cm3); ii) markers of bone turnover - Bone Specific Alkaline Phosphatase (BALP), telopeptide (CTX), Sclerostin and RANK Ligand (RANK-L); iii) serum inflammatory markers including high sensitivity C-reactive Protein (hs-CRP), Interleukin-1ß (IL-1ß). interleukin-6 (IL-6), tumor necrosis factor - alpha (TNF-alpha), erythrocyte sedimentation rate (ESR); and, iv) lipid profile; low density lipoprotein cholesterol (LDL), high density lipoprotein cholesterol (HDL), triglycerides, and total cholesterol Clinical Implications: Should rosuvastatin prove to be safe and efficacious for reducing endocrine metabolic disease risk for adults with chronic SCI, the results will advance the health of people with SCI by reducing the frequency and severity of heart disease and fracture as they age, with a single intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18-60 years)
* Motor complete SCI (C1-T10 AIS A/B)
* 2 years post-injury
* Have a telephone, and ability to attend the study visits
* Able to take oral medications and swallow independently
* Can provide free and informed consent
* Ability to understand instructions in English
* May report current use of oral alendronate 10mg daily or 70mg weekly or risedronate 5mg daily, 30mg weekly or 150mg monthly

Exclusion Criteria:

These criteria are intended to exclude those in whom; Rosuvastatin would be unsafe, DXA/pQCT measurement or biomarker assessment would be invalid, or in whom other co-morbid health conditions may confound the study results. Exclusion criteria include:

* Current and/or one year prior to enrolment treatment with any statin such as atorvastatin, fluvastatin, lovastatin, pitavastatin, pravastatin, simvastatin and rosuvastatin.
* Current treatment with IV bisphosphonate, denosumab, recombinant PTH, ovarian hormone therapy, an oral contraceptive, Immunosuppressants (Including Cyclosporine) and fusidic acid.
* Known allergy to Rosuvastatin, lactose powder, CoQ10, calcium carbonate, vitamin D2 and vitamin D3, or any other ingredient found in rosuvastatin, placebo or study supplements.
* History of Paget's disease, osteomalacia, steroid induced osteoporosis, or untreated parathyroid or untreated thyroid disease.
* Subjects with history of stage 4 chronic kidney disease. (124)
* Current Weight ≥136 kg.
* Bilateral knee region metal implants (hardware), history of bilateral knee region contracture >30 degrees, fracture or any other bilateral knee region pathology which would preclude accurate DXA assessment of one limb.
* Post-menopausal women (absence of menses for a minimum of 1 year).
* Women with amenorrhea due to bilateral surgical removal of the ovaries and/or uterus (women with amenorrhea due to spinal cord injury are able to participate).
* Pregnancy or lactation.
* Female of child-bearing potential who is engaged in active heterosexual relations and is not using appropriate birth control methods. Appropriate methods of birth control will include: surgical sterilization at least 6 months prior to using study drug or sexual activity restricted to a vasectomized partner, barrier contraception with a condom or diaphragm in conjunction with spermicidal gel in use at least 30 days prior to using study drug OR sexual abstinence as a lifestyle.
* History of liver disease or abnormal Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT), ≥1.5 times the upper limit of the normal reference range at enrolment.
* History of symptomatic hypocalcemia or hypophosphatemia.
* Concurrent treatment with prednisone (>7.5mg/day for 90 days).
* Vitamin D deficiency (Serum Vitamin D level <75nmol/L) after completing 8 to 12 weeks of treatment for Vitamin D deficiency as per the Vitamin D correction protocol (Appendix Page 1).
* History of heart attack or stroke.
* Untreated hypertension defined as: elevated BP above (135/85mmHg) assessed with an automated blood pressure cuff at 3 distinct time points in a 7-10 day period.(125, 126)
* Current alcohol or street drug abuse.
* Any illness or condition interfering with the trial conduct or subject safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in areal BMD of the knee region | Baseline and 12 months (or study completion)
  Dual Xray Absorptiometry (DXA) Assessment of areal bone mineral density (aBMD) of the knee region

SECONDARY OUTCOMES:
Change from Baseline in Low density lipoprotein cholesterol (LDL) | Baseline and 12 months (or study completion)
  Serum assessment of LDL
Change from Baseline in high density lipoprotein cholesterol (HDL) | Baseline and 12 months (or study completion)
  Serum assessment of HDL
Change from Baseline in triglycerides (TG) | Baseline and 12 months (or study completion)
  Serum assessment of TG
Change from Baseline in total cholesterol | Baseline and 12 months (or study completion)
  Serum assessment of cholesterol
Change from Baseline in High sensitivity C-reactive Protein (hsCRP) | Baseline and 12 months (or study completion)
  Serum assessment of hsCRP
Change from Baseline in Interleukin-1ß (IL-1ß) | Baseline and 12 months (or study completion)
  Serum assessment of IL-1ß
Change from Baseline in interleukin-6 (IL-6) | Baseline and 12 months (or study completion)
  Serum assessment of IL-6
Change from Baseline in tumor necrosis factor - alpha (TNF-alpha) | Baseline and 12 months (or study completion)
  Serum assessment of TNF-alpha
Change from Baseline in erythrocyte sedimentation rate (ESR) | Baseline and 12 months (or study completion)
  Serum assessment of ESR
Change from Baseline in Bone Specific Alkaline Phosphatase (BALP) | Baseline, 6 months and 12 months (or study completion)
  Serum assessment of BALP
Change from Baseline in C-telopeptide (CTX) | Baseline, 6 months and 12 months (or study completion)
  Serum assessment of CTX
Change from Baseline in Sclerostin | Baseline, 6 months and 12 months (or study completion)
  Serum assessment of Sclerostin
Change from Baseline in RANK Ligand (RANK-L) | Baseline, 6 months and 12 months (or study completion)
  Serum assessment of RANK-L
Change from Baseline in volumetric BMD of the tibia (pQCT) | Baseline and 12 months (or study completion)
  Peripheral Quantitative Computed Tomography (pQCT) assessment - Toronto Site Only
Change from Baseline in volumetric BMD of the tibia (HR-pQCT) | Baseline and 12 months (or study completion)
  High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT) assessment - Toronto Site Only

OTHER OUTCOMES:
Changes in visceral adipose tissue | Baseline and 12 months (or study completion)
  Whole Body DXA assessment of body composition
Changes in lean mass | Baseline and 12 months (or study completion)
  Whole Body DXA assessment of body composition
Changes in aortic arterial stiffness | Baseline and 12 months (or study completion)
  Assessment of Aortic Pulse Wave Velocity (aPWV)

CONTACTS AND LOCATIONS:
Overall Officials: B. Catharine Craven, BA, MD, FRCPC, MSc, Principal Investigator — Toronto Rehabilitation Institute - UHN
Locations (2):
- University Of Miami Miller School of Medicine, Miami, Florida, United States
- University Health Network - Toronto Rehab Lyndhurst Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No